CLINICAL TRIAL: NCT05175196
Title: Microengineered Lollipop for Patient-Centric Saliva Collection
Brief Title: CandyCollect Strep Throat Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-1427; A536756 (Other: UW Madison); Protocol Version 2/28/2025 (Other: UW Madison); SMPH\PEDIATRICS\INFECT DIS (Other: UW Madison); R21AI166120 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-04

CONDITIONS: Group A Streptococcal Infection
Keywords: saliva collection; diagnosis; pediatric
MeSH Terms: conditions — Streptococcal Infections; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pediatric Participants with GAS (Experimental): Children age 5-17 years old diagnosed via standard Rapid Antigen Detection Test with acute pharyngitis caused by Group A Streptococcus (GAS), along with their parent or legal guardian (aka "caregiver").
  Interventions: Diagnostic Test: CandyCollect; Diagnostic Test: Lollipop Swab

INTERVENTIONS:
Diagnostic Test: CandyCollect — The CandyCollect device is a novel, micro-engineered, lollipop-inspired platform. It has functionalized open microchannels for pathogen capture and concentration. It also has time-controlled flavoring release to make the platform more patient-centric.
Diagnostic Test: Lollipop Swab — The "lollipop" swab is a typical swab that would be used to obtain routine pharyngeal samples. Child participants are instructed to suck on the swab for 10 seconds, as they would suck on a lollipop. Participant will be asked to take this test twice.

SUMMARY:
This study will enroll children ages 5-17 who test positive for Group A Streptococcus (GAS) at a single clinic visit lasting approximately 30-60 minutes. The primary aim of this study is to assess the accuracy and feasibility of the CandyCollect platform to capture and detect GAS. The investigators hypothesize that the CandyCollect platform is non-inferior to gold-standard rapid antigen detection testing for GAS.

DETAILED DESCRIPTION:
The rationale for this study is to demonstrate the potential of the CandyCollect platform for acquisition of samples from children in the clinic. With deliberate design to maximize collection performance from saliva sampling, the investigators long-term vision is that the CandyCollect platform will achieve better sensitivity and specificity than can be obtained with current biospecimen collection techniques, while providing a platform that is preferred by patients and usable in home settings. Ultimately, the CandyCollect has the potential to make saliva sampling a new gold standard for respiratory disease diagnostics and prevent the discomfort associated with a pharyngeal swab.

The Theberge Lab at the University of Washington that is developing CandyCollect is using data collected throughout the study to iterate the engineering of the device. As such, analyses were performed after Cohort 1 (n=30 dyad completers), and in line with the iterative nature of this study, the study team adjusted the study design to further inform the engineering of the device. For Cohort 2, which will also target n=30 dyad completers, the study team will still administer surveys to the child and caregiver and collect 4 saliva samples from each child. Cohort 3 will target n= 30 dyad completers, and the study team will administer surveys and collect 5 saliva samples from each child.

Intervention:

* Cohort 1: Pediatric participants diagnosed with GAS via rapid antigen detection test (RADT) will be asked to suck on a swab for 10 seconds, like sucking on a lollipop. They will then be asked to suck on a candy lollipop that will collect their saliva. Participants will do each type of saliva collection twice-two swabs, then two lollipops. Afterwards, participants (both pediatric and caregiver) will fill out a short survey asking about their feelings and opinions about the different types of tests.
* Cohort 2: Pediatric participants diagnosed with GAS via rapid antigen detection test (RADT) will be asked to suck on four CandyCollect devices and one lollipop swab. The CandyCollect devices will be designed such that one will take 10 seconds to obtain, one will take 30 seconds to obtain; and two will each take 1 minute to obtain; participants will be instructed to suck on the CandyCollect device for these durations. Afterwards, participants (both pediatric and caregiver) will fill out a short survey asking about their feelings and opinions about the different types of tests.
* Cohort 3: Pediatric participants diagnosed with GAS via rapid antigen detection test (RADT) children will use the first four CandyCollect devices for 1 minute and the fifth CandyCollect device until it dissolves (about 1.5 - 3.5 minutes). They will also use 1 lollipop swab. [Cohort 3 is not funded by NIH]

Specific aims:

* Aim 1: The primary aim of this study is to assess the efficacy of the CandyCollect platform to capture and detect GAS in a small scale clinical study. The investigators will compare results of the CandyCollect sampling with both the RADT, which is the current gold standard, as well as a lollipop swab.
* Aim 2: The secondary aim of this study is to evaluate the usability of the CandyCollect device by surveying pediatric participant and parent experience, acceptance of the collection technique, and their willingness to perform the test at home.

Hypotheses to be tested:

* Aim 1: The CandyCollect platform is non-inferior to gold-standard RADT for GAS.
* Aim 2: Pediatric participants and their parent/legal guardians will have a more positive experience with the CandyCollect than the RADT throat swab or the lollipop swab, and they will be willing to do the CandyCollect at home.

ELIGIBILITY:
Inclusion Criteria:

* Child age 5-17 years old
* Diagnosis of acute pharyngitis caused by GAS
* A positive RADT swab in clinic
* Able to assent and complete surveys in English

Exclusion Criteria:

* Unable to suck on a swab or CandyCollect
* Previous participation in this study
* Self-reported sensitivity to sugar-free products

Inclusion for Caregiver Participants:

* Parent or legal guardian able to provide consent for child participant
* Physically present at the clinic with the child
* Able consent and complete surveys in English

Exclusion for Caregiver Participants:

* Does not meet inclusion criteria

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of test results positive for GAS | day 1 (up to 40 minutes)
  The primary aim of this study is to assess the efficacy of the CandyCollect platform to capture and detect Group A Streptococcus (GAS) in a small scale clinical study. The investigators will compare results of the CandyCollect sampling and a lollipop swab test to the rapid antigen detection test (RADT).

SECONDARY OUTCOMES:
Caregiver Experience Score (Bad/Good) | day 1 (up to 40 minutes)
  The secondary aim of this study is to evaluate the usability of the CandyCollect device by surveying participant experience with the throat swab, lollipop swab, and CandyCollect. Caregivers will be asked to rate their experiences on a scale of -5 (bad) to 5 (good). Mean scores for each feeling for each test will be reported.
Caregiver Experience Score (Pleasant/Unpleasant) | day 1 (up to 40 minutes)
  The secondary aim of this study is to evaluate the usability of the CandyCollect device by surveying participant experience with the throat swab, lollipop swab, and CandyCollect. Caregivers will be asked to rate their experiences on a scale of 1 (pleasant) to 7 (unpleasant). Mean scores for each feeling for each test will be reported.
Caregiver Sample Collection Preference | day 1 (up to 40 minutes)
  The acceptance of the CandyCollect device relative to other sample collection methods will be measured by surveying preferred sample collection method for their child if they needed another test next week, which method they preferred, which method was most suitable for children in general, and which method was least invasive. Count of Caregivers for each question for each sample collection method will be reported.
Number of Caregivers Willing to Have Their Child Perform the CandyCollect at Home | day 1 (up to 40 minutes)
  Acceptability of the CandyCollect device will be in part measured by Caregiver willingness to perform the test at home.
Pediatric Participant Wong-Baker FACES Pain Score for Each Sample Collection Method | day 1 (up to 40 minutes)
  Pediatric participants will be surveyed with the Wong-Baker FACES Pain Rating Scale for their experience with the throat swab, lollipop swab, and CandyCollect. Scores range from 1-10, where higher scores indicate increased pain.
Pediatric Participant Yummy / Yucky Score for Each Sample Collection Method | day 1 (up to 40 minutes)
  Pediatric participants will be surveyed with Yummy to Yucky Scale for their experience with the throat swab, lollipop swab, and CandyCollect. Scores range from 1-5, where higher scores indicate worse experience.
Pediatric Participant Sample Collection Preference | day 1 (up to 40 minutes)
  Pediatric participants will be asked with sample collection method they prefer: throat swab, lollipop swab, or CandyCollect.
Number of Pediatric Participants Willing to do the CandyCollect at Home | day 1 (up to 40 minutes)
  Acceptability of the intervention will be in part measured by asking pediatric participants if they are willing to do the CandyCollect at home.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory DeMuri, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No